CLINICAL TRIAL: NCT05166330
Title: Comparison of Different Ratios of Propofol-ketamine Admixture in Rapid-sequence Induction of Anesthesia for Emergency Laparotomy: a Randomized Controlled Trial
Brief Title: Two Ratios of Propofol-ketamine Admixture for Rapid-sequence Induction Anesthesia for Emergency Laparotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-450-2021
Record Dates: First submitted 2021-11-24; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Hypotension; Induction of Anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketofol 1:1 (Active Comparator): 0.15-0.2 mL/kg from of 5 mg/mL propofol and 5 mg/mL ketamine mixture
  Interventions: Drug: Ketofol equal ratio
- ketofol 1:3 (Active Comparator): 0.15-0.2 mL/kg from of 7.5 mg/mL propofol and 2.5 mg/mL ketamine mixture
  Interventions: Drug: Ketofol 1:3 ratio

INTERVENTIONS:
Drug: Ketofol equal ratio — 5mg/ml10 mL propofol (100 mg) will be mixed with 2 mL ketamine (100 mg) and then diluted to a total volume of 20 mL to have a final concentration of 5 mg/mL propofol and 5 mg/mL ketamine
  Arms: ketofol 1:1
Drug: Ketofol 1:3 ratio — 15 mL propofol (150 mg) will be mixed with 1 mL ketamine (50 mg) and then diluted to a total volume of 20 mL to have a final concentration of 7.5 mg/mL propofol and 2.5 mg/mL ketamine).
  Arms: ketofol 1:3

SUMMARY:
Hypotension during anesthesia is associated with serious organ failure and death. The most critical period for intraoperative hypotension is the postinduction period during which, one-third of intraoperative hypotension occurs. Post-induction hypotension has many contributing factors; however, it is closely related to anesthetic drugs. Therefore, manipulation of induction agents makes post-induction hypotension likely preventable. Emergency laparotomy is a critical category of surgery whose patients are usually hemodynamically compromised and prone to post-induction hypotension; furthermore, these patients are usually at high risk of aspiration of gastric contents and require rapid-sequence induction of anesthesia and optimum intubating conditions. Thus, induction of anesthesia for emergency laparotomy requires meticulous balance between achievement of adequate hypnosis and maintenance of stable blood pressure.

Propofol is the commonest hypnotic agent worldwide. However, it is usually associated with hypotension especially in compromised patients. Ketamine produces dissociative anesthesia and sympathetic stimulation which provides more stable hemodynamic profile; however, ketamine is not widely used as a routine hypnotic because it produces psychomimetic effects such as delirium and emergence agitation. Nevertheless, ketamine still has a role in induction of anesthesia in patients with shock and during procedural sedation. Ketamine is also used as analgesic adjuvant during general anesthesia.

Propofol/ketamine admixture (ketofol) was introduced in anesthetic practice aiming to compensate the side effects of the two drugs and to provide, consequently, the desired balance between adequate hypnosis and hemodynamic stability. Ketofol is currently used with a diversity in the ratio between the two drugs which ranges between 1:1 and 1:10 between ketamine and propofol. Despite its frequent use in sedation and complete anesthesia, most of the available literature for comparisons of different ketofol mixtures was restricted to procedural sedation whose results are not applicable in induction of anesthesia due to the different desirable level of hypnosis and recovery. Therefore, the best combination of the two components of ketofol for induction of anesthesia is unknown

DETAILED DESCRIPTION:
Preoperatively, a trained anesthetist will assess the patients regarding the fasting hours, medical history, medications, laboratory investigation, as well as the patient's airway.

In the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and routine pre-medications (dexamethasone 4 mg as 0.5 mg/ml slow I.V injection) will be administrated. Baseline preoperative blood pressure will be recorded in the supine position as average of 3 readings with difference less than 10% in the systolic blood pressure.

After 3-minutes preoxygenation, patients in the two groups will receive 1 mg/kg lidocaine (in a separate syringe) plus 0.15-0.2 mL/kg from the prepared mixture. This regimen will provide a dose of 1 mg/kg propofol + 1 mg/kg ketamine in the ketofol-1:1 group and 1.5 mg/kg propofol + 0.5 mg/kg ketamine in the ketofol-1:3 group.

Clinical loss of consciousness (defined as no response to auditory command and the disappearance of a patient's eyelash reflex). After loss of consciousness, succinylcholine 1 mg/kg will be administered over 5 seconds, and tracheal intubation will be done through direct laryngoscopy after 60 seconds.

The intubation conditions will be graded by the same anesthetist who performed intubation as excellent, good, or poor for :ease of laryngoscopy, Vocal cord position, Reaction to insertion of the tracheal tube and cuff inflation (Diaphragmatic movement/coughing) Excellent, all criteria excellent; good, all criteria either excellent or good; poor, presence of a single criterion graded as poor.

When the trachea is intubated, mechanical ventilation will be applied to obtain SpO2 > 95% and end-tidal CO2 between 30-40 mmHg and anesthesia will be maintained by isoflurane. Atracurium will be administered after patient recovery from succinylcholine at a dose of 0.5 mg/Kg. Atracurium increments of 10 mg will be administered every 20 min for maintenance of muscle relaxation.

Any episode of hypotension (defined as mean arterial pressure [MAP] <70 mmHg) will be managed by 5 mcg norepinephrine (which will be repeated if hypotension persists for 2 minutes).

If hypertension or tachycardia occurred (defined as MAP or heart rate >120% of baseline), it will be managed by IV 0.5 mg/kg propofol.

After skin incision, hemodynamic and anesthetic management will be according to the attending anesthetist discretion.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-65 years),
* American society of anesthesiologist I-III,
* scheduled for emergency laparotomy under general anesthesia

Exclusion Criteria:

* history of difficult intubation,
* abnormal airway examination,
* cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions),
* patients on angiotensin converting enzyme inhibitors and angiotensin receptor blockers medications,
* patients with uncontrolled hypertension,
* patient with allergy of any of the study drugs
* Patients on vasopressor infusion,
* patients with high shock index (heart rate / systolic blood pressure >1),
* body mass index > 35 kg/m2, increased intracranial tension
* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
norepinephrine dose | 1 minute after induction of anesthesia until 15-minutes after induction
  microgram

SECONDARY OUTCOMES:
postinduction hypotension | 1 minute after induction of anesthesia until 15-minutes after induction
  mean arterial pressure <70 mmHg
severe postinduction hypotension | 1 minute after induction of anesthesia until 15-minutes after induction
  mean arterial pressure <60 mmHg
postinduction hypertension | 1 minute after induction of anesthesia until 15-minutes after induction
  mean arterial pressure >120% baseline
intubation condition | 60 seconds after induction of anesthesia to 180 seconds after induction
  *Excellent, all criteria excellent; good, all criteria either excellent or good; poor, presence of a single criterion graded as poor
  * Ease of laryngoscopy Excellent: Easy: jaw relaxed, no resistance to blade insertion Good : Fair: jaw not fully relaxed, slight resistance to blade insertion Poor: Difficult: poor jaw relaxation, active resistance of the patient to laryngoscopy
  * Vocal cord position Excellent: Abducted Good : Intermediate/moving Poor: Closed
  * Reaction to insertion of the tracheal tube and cuff inflation (Diaphragmatic movement/coughing) Excellent: None Good: Diaphragm/slight: One to two weak contractions or movement for less than 5 s. Poor: Sustained/ Vigorous: More than two contractions and/or movement for longer than 5 s.
total propofol dose | 0 second after induction of anesthesia to 180 seconds after induction
  mg

OTHER OUTCOMES:
mean arterial pressure | 1-minte before the induction, immediately after induction, immediately after intubation, then every 2-minutes for 15-minutes after induction
  mmHg
heart rate | 1-minte before the induction, immediately after induction, immediately after intubation, then every 2-minutes for 15-minutes after induction
  beat per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
will be provided upon reasonable request

REFERENCES:
- [Derived] Elsherbiny M, Hasanin A, Kasem S, Abouzeid M, Mostafa M, Fouad A, Abdelwahab Y. Comparison of different ratios of propofol-ketamine admixture in rapid-sequence induction of anesthesia for emergency laparotomy: a randomized controlled trial. BMC Anesthesiol. 2023 Oct 3;23(1):329. doi: 10.1186/s12871-023-02292-w. PMID 37789329